CLINICAL TRIAL: NCT02274142
Title: Minimally Invasive Restorations in Primary Molars Using Encapsulated ou Hand-mixed Glass Ionomer Cement: Clinical Trial With 24 Months of Follow-up
Brief Title: Primary Molars Restorations With Encapsulated or Hand-Mixed Glass Ionomer: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MICARDEC
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
Keywords: dentinal caries; occlusal; occluso-proximal
MeSH Terms: conditions — Dental Caries; Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restorations with Encapsulated material (Experimental): Restorations performed with encapsulated glass ionomer cement (EQUIA - GC Corp). Capsules with glass ionomer will be activated and applied after selective carious tissue removal in primary molars.
  Interventions: Procedure: Restoration with Encapsulated material; Device: Encapsulated glass ionomer cement (EQUIA - GC Corp).
- Restorations with Hand-Mixed material (Active Comparator): Restorations will be performed with hand-mixed glass ionomer cement (Fuji IX - GC Corp) after selective carious tissue removal in primary molars.
  Interventions: Procedure: Restoration with hand-mixed material; Device: powder-liquid glass ionomer cement (Fuji IX - GC Corp)

INTERVENTIONS:
Procedure: Restoration with hand-mixed material — restoration with hand-mixed glass ionomer cement
  Other Names: Minimally invasive restoration
  Arms: Restorations with Hand-Mixed material
Procedure: Restoration with Encapsulated material — restoration with encapsulated ionomer cement
  Arms: Restorations with Encapsulated material
Device: Encapsulated glass ionomer cement (EQUIA - GC Corp).
  Arms: Restorations with Encapsulated material
Device: powder-liquid glass ionomer cement (Fuji IX - GC Corp)
  Arms: Restorations with Hand-Mixed material

SUMMARY:
The aim of this RCT is to evaluate the survival of different glass ionomer cement in minimally invasive restorations, with different handling characteristics: hand-mixed versus encapsulated.

DETAILED DESCRIPTION:
Detailed Description: This study was approved by the research ethics committee of the School of Dentistry (University of São Paulo, Brazil) and written informed consent will be obtained from the parents or legal guardians. The sample size was calculated based on the data obtained in a systematic review, which reported average longevity of 78% after 2 years of follow up (mean survival of occlusal and occlusoproximal surfaces). The minimum difference of 15% in the success rate between the control and treatment groups after 2 years of follow-up, with and α of 5% and power (strength) of 80% using paired test. As more than one tooth per children might be included, we must add a 20% for clustering. Adding 20% for possible losses the final estimate is 116 teeth per group, reaching a final sample of 232 teeth.

Inclusion Criteria:

* Children who have sought treatment in the School of Dentistry, University of Sao Paulo;
* Children between 3 and 10 years old without systemic diseases;
* Children presenting at least one dentin caries cavity in primary teeth (occlusal or oclusoproximal) with no signs of pulp involvement.

Exclusion Criteria:

* Children whose parents did not agree to participate in the study;
* Children with behavioural issues at the initial exam or who did not assent to participate in the study.

Implementation:

All the occlusal and occlusoproximal restorations will be performed by two operators on the dental chair. The operators will be assisted by another dentist, who will be previously trained to mix the GIC according to the manufacturers' protocol. The children will be randomly assigned into two groups: Hand-mixed and encapsulated materials.

Treatment procedure:

The restorative technique will be performed according to the Minimal Intervention Dentistry. No local anaesthesia will be used during treatment. Rotary instruments can be used to open or to expand the cavity opening, removing only enamel. Infected carious dentin will be removed with hand instruments. The use of hand instruments on the dentin surface results in a smear layer and need to be removed by the use of dentine conditioner. The liquid component of the hand-mixed powder-liquid GIC, containing the acid component, will be used and saliva isolation will be done with cotton wool rolls. The cavities will be restored with one of the two GIC brands: Fuji IX (GC Europe, Leuven, BE) and EQUIA (GC Europe, Leuven, BE). A thin layer of petroleum jelly will be rubbed over the index finger and the restoration will be pressed for 20 seconds. The material will include sealing pits and the fissure. After preparing for a balanced occlusion, a new layer of petroleum jelly will be applied to the GIC restoration. The amount of GIC used, element number, cavity dimension and dmft will be recorded. The duration of the restorative procedure will be recorded with a stopwatch. The participating children will be instructed not to eat for one hour after the restoration is placed.

Evaluation:

The success of the restorations will be evaluated after 6 months according to the Frencken and Holmgren criteria for occlusal surfaces, and modified version of Roeleveld et al. (2006) criteria for occlusoproximal surfaces. A restoration will be considered as 'failure' when there is a defect in the filling when secondary caries is observed, when the restoration is not present or when the pulp is inflamed. When the restoration is still present or a slight defect is observed, it will be considered as 'success'. When the tooth is unavailable for evaluation, it will be censored. All evaluations will be carried out by two independent evaluators, who did not restore the cavities, trained and calibrated by a benchmark.

Estimation of cost-effectiveness:

The material cost (GICs) will be estimated per restoration. The average cost per restoration will be estimated. Costs of equipment, autoclave and hand instruments, disposables (hand gloves, face masks, cotton wool rolls), articulating paper and petroleum jelly used for the restorations are equal for both GIC groups and will be excluded. There will be no labour costs for the operators.

ELIGIBILITY:
Inclusion criteria:

* Children who have sought treatment in the School of Dentistry, University of Sao Paulo;
* Children between 3 and 10 years old without systemic diseases;
* Children presenting at least one dentin caries cavity in primary teeth (occlusal or oclusoproximal) with no signs of pulp involvement.

Exclusion Criteria:

* Children whose parents did not agree to participate in the study;
* Children with behavioural issues at the initial exam or who did not assent to participate in the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Restorations survival | 24 months
  The survival of restorations will be evaluated over 24 months according to the Frencken and Holmgren (1999) index for occlusal cavities and Roeleveld (2006) for occlusoproximal cavities.

SECONDARY OUTCOMES:
Cost-Effectiveness | 24 months
  Cost-effectiveness will be measured according to each restoration performed and the cost of all reinterventions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Raggio, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Oliveira RC, Camargo LB, Novaes TF, Pontes LRA, Olegario IC, Gimenez T, Passaro AL, Tedesco TK, Braga MM, Mendes FM, Raggio DP. Survival rate of primary molar restorations is not influenced by hand mixed or encapsulated GIC: 24 months RCT. BMC Oral Health. 2021 Jul 23;21(1):371. doi: 10.1186/s12903-021-01710-0. PMID 34301217